CLINICAL TRIAL: NCT02546622
Title: A Longitudinal, Observational Study of Previously Treated Hemophilia Patients Switching Factor Replacement Products
Brief Title: ATHN 2: Factor Switching Study
Status: Completed | Type: Observational
Sponsor: American Thrombosis and Hemostasis Network (Network)
Collaborators: Shire (Industry); CSL Behring (Industry); Bioverativ Therapeutics Inc. (Industry); Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: ATHN 2
Record Dates: First submitted 2015-09-09; First posted 2015-09-11 (Estimated); Last update posted 2021-12-09 (Actual); Status verified 2020-08

CONDITIONS: Hemophilia
Keywords: Factor; Coagulation; Inhibitor; HTC; Bleeding
MeSH Terms: conditions — Hemophilia A; Thrombosis; Hemorrhage | interventions — factor VIII-Fc fusion protein; recombinant factor VIII N8; BAX 855; Factor VIII; F8 protein, human; factor IX Fc fusion protein; albutrepenonacog alfa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: None Retained — Plasma drawn at baseline, after 10 Exposure Days, after 50 Exposure Days, and at study end (1 year). If inhibitor suspected, sample will be drawn and tested locally, and within 2 weeks of first positive inhibitor, a confirmatory sample will be drawn and sent to CDC. Patients may be co-enrolled in other ATHN studies such as My Life Our Future, will performs genotype Samples may be linked in patient who have authorized
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Arm A Prospective: Patients who are switching to a new Factor VIII and Factor IX Replacement Product for Hemophilia A and B which was FDA approved after January 1, 2013.
  These patients will be followed prospectively for up to 1 year.
  Interventions: Biological: Factor VIII Replacement Products for Hemophilia which were FDA approved after January 1, 2013; Biological: Factor IX Replacement Products for Hemophilia which were FDA approved after January 1, 2013
- Arm B Retrospective: Patients who have recently switched to a new Factor VIII and Factor IX Replacement Product for Hemophilia A and B which was FDA approved after January 1, 2013.
  Patients must have switched products within the past 50 weeks at the time of enrollment.
  These patients will be assessed retrospectively and/or followed prospectively for up to 1 year.
  Interventions: Biological: Factor VIII Replacement Products for Hemophilia which were FDA approved after January 1, 2013; Biological: Factor IX Replacement Products for Hemophilia which were FDA approved after January 1, 2013

INTERVENTIONS:
Biological: Factor VIII Replacement Products for Hemophilia which were FDA approved after January 1, 2013 — Prophylaxis for prevention of bleeding, various regimens.
  Other Names: Eloctate®; NovoEight®; Adynovate®; Nuwiq®; Afstyla®; Kovaltry®
Biological: Factor IX Replacement Products for Hemophilia which were FDA approved after January 1, 2013 — Prophylaxis for prevention of bleeding, various regimens.
  Other Names: Alprolix®; Rixubis®; IXinity®; Idelvion®; Rebinyn®

SUMMARY:
This is a longitudinal, observational study of patients with Hemophilia A or B who are planning to switch to a newly approved coagulation factor replacement product, or who have recently switched factor products. The study will follow each patient for up to 1 year. Patients will be recruited at Hemophilia Treatment Centers (HTC) which are ATHN-affiliates. The primary outcome being studied is the development of inhibitor (i.e., antibodies to factor) at 1 year or 50 exposure days, whichever comes first.

The study will be conducted at approximately 30 HTCs, with a planned enrollment of 600 patients.The entire study duration is projected to be approximately 6 years.

In addition, optional substudies will be included for some products, as "Product-Specific Modules". These will be questionnaires to collect data for subjects receiving selected Factor products. For example, subjects receiving Kovaltry will be approached to participate in the 'Kovaltry Product-Specific Module'; subjects receiving Adynovate will be approached to participate in the 'Adynovate Product-Specific Module'. Questions will be related to product use, perceptions of product use, and other post-marketing consumer data.

DETAILED DESCRIPTION:
This non-interventional, minimal risk cohort study will enroll patients with Hemophilia A or B who are planning or have recently switched to a new Factor product. The study will have 2 Arms, prospective and retrospective. The Prospective Arm will enroll patients who plan to switch to a new factor. The Retrospective Arm will enroll patients who have recently switched to a new factor (within the previous 50 weeks). Patient will be seen at baseline and for up to 4 additional visits, and quarterly follow-up by phone. Required study visits will be planned to coincide with routine follow-up visits whenever possible.

Please note that Factor Replacement Products are not being provided by the study.

The primary objective is to assess and characterize the rate of inhibitor development within one (1) year or fifty (50) exposure days, whichever is first, after switching clotting factor replacement products in previously treated patients (PTPs) with hemophilia A or B.

Data collected will include eligibility, demographics, medical history, hemophilia history (clotting history, product history, genotype and family history), inhibitor history, co-morbidities at baseline (i.e., HIV, Hepatitis C.), detailed clotting factor replacement product(s) usage and switching plan, and reasons for switching factor products. Also targeted physical exams will be performed at baseline and during follow-up, and targeted concomitant medication data will be collected. Data collection will also include patient-reported outcome(s) after 1 year, bleeding events, surgeries, laboratory Inhibitor testing and details regarding testing methodology, pharmacokinetic (PK) data (if known), new diagnoses, and co-morbidities (targeted), Safety/Adverse Events using European Union Hemophilia Safety Surveillance (EUHASS) definitions.

This study will evolve to include any newly approved (since January 2013) factors as they come to market. Cohorts will be defined by the brand/type of new clotting factor replacement product approved after January 1, 2013. The current list of specific new Factor VIII replacement products include Eloctate® (Bioverativ) and NovoEight® (NovoNordisk); Factor IX replacement products include Alprolix® (Bioverativ), Rixubis® (Baxalta), and IXinity® (Emergent Biosolutions). Others are both now available and imminent and include: Adynovate®, Idelvion®, Afstyla®, Kovaltry® and Jivi®.

The over-arching rationale for this protocol is that a pragmatic study which is consistent with real world practices across a wide range of patients that is not principally tied to a particular manufacturer or product may be of great advantage to the entire hemophilia community.

Study Duration

* Subjects on prophylaxis will be followed on study for up to 1 year. Each subject will be seen during a study visit or contacted by telephone at least once every 3 months (i.e., quarterly). Patients may participate for multiple 'cycles', if they switch factor products more than once while the study is actively recruiting.

Treatment regimen will be at the discretion of the subject's hemophilia caregivers. No treatment is being provided by the study.

* Substudies A number of substudies are planned with pharmaceutical sponsors to collect information from patients about their products' use. Participation in these optional substudies (product-specific modules) will be planned to coincide with study visits. These modules will collect information from subjects about their perception and use of factor use/treatment, physical activity levels and other general health questions. These data will be collected via questionnaire, primarily via phone.

Concomitant and Excluded Therapies

* Immune tolerance therapy is excluded on study. This includes immunosuppressive treatments used to eradicate inhibitors. Steroid treatments for allergic disorders and asthma, are allowed.

Data Collection System

* All data collected will be entered into electronic case report forms (eCRFs) within the secure ATHN Study Manager system. Subject Identifiers (IDs) will be generated in Clinical Manager.
* Reimbursement will be managed by each participating HTC. Most study centers will reimburse study subjects for travel and parking, but this varies by center.

ELIGIBILITY:
Inclusion Criteria

* Moderate or Severe Congenital Hemophilia A or B (FVIII or FIX clotting activity less than or equal to 5% of normal).
* Able to give informed consent (by patient or parent/authorized guardian).
* Previously treated with plasma-derived or recombinant clotting factor replacement products with at least 50 exposure days (as assessed either from direct clinical records in children under age 5, or by clinical history of dosing in older patients). For Arm B being enrolled retrospectively, this previous treatment must be prior to product switch under study.
* Planning to switch, or recently switched within the previous 50 weeks, to a new brand or type of replacement factor VIII or IX, FDA approved after January 1, 2013.
* Arm B only: Negative inhibitor screen within the last 6 months prior to switching.

Note: History of prior transient inhibitor or inhibitor eradicated by immune tolerance induction (ITI) are eligible.

Exclusion Criteria

* Presence of any known bleeding disorder other than hemophilia A or B (i.e., patients with concurrent hemophilia and a second hemostatic defect are NOT eligible). Low Von Willebrand Factor (VWF) without VWF diagnosis are not excluded.
* Presence of an active inhibitor >0.6 BU for factor VIII, > 0.4 BU for factor IX at the time of eligibility assessment. Detection of such an inhibitor at the baseline visit prior to dosing with the new product (Arm A), or after dosing with new factor dosing (Arm B), would result in early termination without other study assessments.
* Currently undergoing ITI.
* Immunosuppressive therapy (cyclophosphamide, mycophenolate, IVIG) within 90 days and Rituximab within 6 months; topical steroid treatments and short course steroids for asthma or allergy allowed.
* Previous participation in Phase I, II or III interventional trials of the factor product being switched to.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will enroll approximately 600 patients with hemophilia who meet the eligibility criteria and are receiving care from one of the ATHN-affiliated Hemophilia Treatment Centers (HTC). There will be 2 arms:
  Arm A (Prospective) will include patients who are switching factor replacement products and will be followed prospectively for up to 1 year.
  Arm B (Retrospective) will include patients who have switched factor replacement products previously (within the past 50 weeks at the time of enrollment). These patients will be assessed retrospectively and/or followed prospectively for up to 1 year.
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2015-09; Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Inhibitor Development | After 50 Exposure Days or 1 Year, whichever comes first
  Inhibitor development is the primary outcome. Subjects will be followed closely and tested at baseline, after 10 Exposure Days and 50 Exposure Days, and/or at 1 year. Specimens will be submitted to local laboratories and evaluated for inhibitor titers, and inhibitors will be confirmed by local laboratories and CDC.

SECONDARY OUTCOMES:
Inhibitor Development | 10 days
  To determine the prospective incidence of inhibitor development after 10 exposure days to a new, novel recombinant factor following a switch from another clotting factor replacement product.
Prevalence of risk factors for inhibitor development | 1 year
  To compare the prevalence of selected risk factors in patients with hemophilia who develop inhibitors following switching to a new product, to those found in subjects who do not develop inhibitors.
Targeted post-marketing approval safety and efficacy data | 1 year
  To collect and summarize targeted post-marketing approval safety and efficacy data for events related to clotting factor replacement products, specifically
  * To collect data on bleeding events following switching factor.
  * To summarize replacement factor product dosing regimens prescribed to the study population.
Platform for additional substudies | 1 year
  To serve as a platform for product-specific questionnaires in cohorts of patients who switch to a particular product.

CONTACTS AND LOCATIONS:
Overall Officials: Ellis J Neufeld, MD, PhD, Principal Investigator — St. Jude Children's Research Hospital; Janna Journeycake, MD, Principal Investigator — Oklahoma Center for Bleeding and Clotting Disorders
Locations (27):
- United States (27):
  - University of California San Diego (UCSD), San Diego, California
  - University of Colorado Denver Hemophilia and Thrombosis Center, Aurora, Colorado
  - Yale Hemophilia Treatment Center, New Haven, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Children's Hospital, Tampa, Florida
  - Children's Healthcare of Atlanta/Emory, Atlanta, Georgia
  - Bleeding and Clotting Disorders Institute, Peoria, Illinois
  - Indiana Hemophilia and Thrombosis Center (IHTC), Indianapolis, Indiana
  - Louisiana Center for Bleeding and Clotting Disorders, New Orleans, Louisiana
  - Maine Hemophilia and Thrombosis Center, Scarborough, Maine
  - Johns Hopkins University Medical Center, Baltimore, Maryland
  - Boston Hemophilia Center at Children's Hospital of Boston, Boston, Massachusetts
  - University of Michigan Hemophilia and Coagulation Disorders Program, Ann Arbor, Michigan
  - Michigan State University Center for Bleeding and Clotting Disorders, East Lansing, Michigan
  - Children's Mercy Hospital, Kansas City, Missouri
  - Dartmouth-Hitchcock Comprehensive Hemophilia and Thrombosis Center, Lebanon, New Hampshire
  - Weill Cornell Medicine, New York, New York
  - Mary M. Gooley Hemophilia Center, Rochester, New York
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia (CHOP), Philadelphia, Pennsylvania
  - Pennsylvania Comprehensive Hemophilia and Thrombophilia Program / Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - The Hemophilia Center of Western Pennsylvania, Pittsburgh, Pennsylvania
  - St Jude Children's Research Hospital, Memphis, Tennessee
  - UTSW Medical Center at Dallas/Children's Medical Center, Dallas, Texas
  - Washington Center for Bleeding Disorders Bloodworks Northwest d/b/a Puget Sound Blood Center, Seattle, Washington
  - Blood Center of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Product-Specific Module data for subjects enrolled in each module will be shared with each sponsor, as appropriate.

REFERENCES:
- [Background] Josephson CD, Abshire T. The new albumin-free recombinant factor VIII concentrates for treatment of hemophilia: do they represent an actual incremental improvement? Clin Adv Hematol Oncol. 2004 Jul;2(7):441-6. PMID 16163220
- [Background] Powell JS. Lasting power of new clotting proteins. Hematology Am Soc Hematol Educ Program. 2014 Dec 5;2014(1):355-63. doi: 10.1182/asheducation-2014.1.355. Epub 2014 Nov 18. PMID 25696879
- [Background] Ragni, MV, Kessler, CM, and Lozier, JN (2009). Clinical aspects and therapy for hemophilia, in Hoffman R, Benz EJ, Shattil, SJ et al eds, Hematology, Basic Principles and Practice, 5th Edition, Churchill Livingstone, Philadelphia, pp 1911-1930.
- [Background] Abshire TC, Brackmann HH, Scharrer I, Hoots K, Gazengel C, Powell JS, Gorina E, Kellermann E, Vosburgh E. Sucrose formulated recombinant human antihemophilic factor VIII is safe and efficacious for treatment of hemophilia A in home therapy--International Kogenate-FS Study Group. Thromb Haemost. 2000 Jun;83(6):811-6. PMID 10896230
- [Background] Mahlangu J, Powell JS, Ragni MV, Chowdary P, Josephson NC, Pabinger I, Hanabusa H, Gupta N, Kulkarni R, Fogarty P, Perry D, Shapiro A, Pasi KJ, Apte S, Nestorov I, Jiang H, Li S, Neelakantan S, Cristiano LM, Goyal J, Sommer JM, Dumont JA, Dodd N, Nugent K, Vigliani G, Luk A, Brennan A, Pierce GF; A-LONG Investigators. Phase 3 study of recombinant factor VIII Fc fusion protein in severe hemophilia A. Blood. 2014 Jan 16;123(3):317-25. doi: 10.1182/blood-2013-10-529974. Epub 2013 Nov 13. PMID 24227821